CLINICAL TRIAL: NCT05209074
Title: A Phase I, Single-Center, Open-Label, Dose De-escalation and Expansion Study Ivosidenib + mFOLFIRINOX in Patients With Resectable Pancreatic Adenocarcinoma
Brief Title: Ivosidenib + mFOLFIRINOX in Patients With Resectable Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7221
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Resectable Pancreatic Cancer
MeSH Terms: interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivosidenib+mFOLFIRINOX (Experimental)
  Interventions: Drug: Ivosidenib; Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: Ivosidenib — Ivosidenibflat dose (250mgor 500mg) daily on day 1 of a 14 day cycle.
Drug: mFOLFIRINOX — mFOLFIRINOX on days 1-3 of a 14-day cycle. Surgical resection after up to ninety (90) days of treatment.

SUMMARY:
This study is a single-arm, phase I trial, up to 16 participants with resectable PDA. The study will examine the efficacy of the mutant IDH1 inhibitor ivosidenib, in conjunction with standard-of-care mFOLFIRINOX in the neoadjuvant setting.

DETAILED DESCRIPTION:
Currently, the standard of care treatment for resectable PDA is surgical resection followed by adjuvant chemotherapy. The use of mFOLFIRINOX in this setting has extended survival significantly. Giving ivosidenibwith mFOLFIRINOXmay work better than treating participants with mFOLFIRINOX alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologicallyor cytologically confirmed diagnosis of pancreatic adenocarcinomaor adenosquamous carcinoma.
* Subjects must have resectable right-sided (head/neck/uncinate) pancreatic cancer based on CT or MRI imaging (pancreas protocol CT of the abdomen and pelvis if possible, MRI with contrast or CT with IV contrast in the absence of a pancreas protocol CT scan, CT of the chest with or without contrast) as determined by the PI or Co-investigators. Participants with contrast allergies may be permitted without contrastscans if approved by the PI or Co-Investigators for safety reasons.
* Male or female subjects age >18 years of age.
* Eastern Cooperative Oncology Group (ECOG) Performance status being 0-1 within 2 weeks of planned start of therapy.
* Subjects must have normal organ and marrow function as defined below within 2 weeks of C1D1:
* Adequate hematologic (white blood cell [WBC] ≥ 3500 cells/mm3; platelet count ≥100,000 cells/mm3; absolute neutrophil count [ANC] ≥1500 cells/mm3; and hemoglobin ≥8 g/dL).
* Adequate hepatic function (aspartate aminotransferase [AST/SGOT] <3x upper normal limit [UNL], alanine aminotransferase [ALT/SGPT] <3x UNL, bilirubin <3x UNL).
* Adequate renal function (serum creatinine <2.0 mg/dL or 177 μmol/L).
* Adequate coagulation ("International Normalized Ratio" or INR must be <1.5) unless on therapeutic blood thinners.
* Screening HgbA1C < 7.0%
* Expected survival ≥3 months in the view of the PI or investigators.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Fertile men must practice effective contraceptive methods (i.e. surgical sterilization, or a condom used with a spermicide) during the study, unless documentation of infertility exists.
* No evidence of clinically significant active infection and no seriousor chronicinfection requiring ongoing antibiotics during the study period.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Inclusion of Women and Minorities
* People of all races and ethnic groups are eligible for participation in this trial.

Exclusion Criteria:

* Subjects under the age of 18yearsof age.
* Subjects with unresectablepancreatic canceror resectableleft-sided (body/tail) pancreatic cancer
* Subjects with endocrine or acinar pancreatic carcinoma.
* Subjects with locally advanced or recurrentpancreatic cancer.
* Subjects with metastatic pancreatic cancer based on imaging.
* Subjects who have received prior radiation therapy, surgical or medical treatment for pancreatic cancer.
* Subjects receiving any other standard or investigational treatment for their PDA.
* Pregnant women or breast feeding women, or women of child-bearing potential not using reliable means of contraception are excluded from this study because the teratogenic or abortifacient effects of ivosidenibis unknown. Because there is an unknown, but potential risk for adverse events in nursinginfants secondary to treatment of the mother with ivosidenib, breastfeeding should be discontinued if the mother is treated withivosidenib. These potential risks may also apply to other agents used in this study.
* Fertile men unwilling to practice contraceptive methods during the study period.
* Subjects with a life expectancy less than 3 months.
* Subjects with a serious medical illness that would potentially increase subjects' risk for toxicity
* Subjects with any active uncontrolled bleeding, and any participants with a bleeding diathesis (e.g., active peptic ulcer disease).
* Subjects with a history of myocardial infarction that is <3 months prior to registration.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure or coronary artery disease, unstable angina pectoris, cardiac arrhythmiarequiring medications that interact with ivosidenib, symptomatic myocardial infarction or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects who are known to be HIV-positive and on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ivosidenib.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) or Recommended Phase 2 dose (RP2D) | Up to 24 months from the start of treatment
  Evaluate by the Bayesian optimal interval (BOIN) strategy to identify the MTD.

SECONDARY OUTCOMES:
RECIST version 1.1 response rates. | Up to 24 weeks from the start of treatment
  Number of participants with the progression-free occurrence.
Major pathologic response rates | Up to 24 weeks from the start of treatment
  Number of participants in whom historical treatment's response rate of 10%
Biochemical response rates | Up to 24 weeks from the start of treatment
  Number of participants with normalization of serum tumor markers during treatment and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: David Bajor, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Zarei M, Hajihassani O, Hue JJ, Graor HJ, Rothermel LD, Winter JM. Targeting wild-type IDH1 enhances chemosensitivity in pancreatic cancer. bioRxiv [Preprint]. 2023 Mar 29:2023.03.29.534596. doi: 10.1101/2023.03.29.534596. PMID 37034685